CLINICAL TRIAL: NCT06181175
Title: Valutazione Dell'Efficacia Del Trattamento Dell'Ipertrofia Prostatica Benigna Con Serenoa Repens Estratta Con CO2 + PEA (Palmitoilethanolamide) in Monoterapia o in Combinazione Alla Tamsulosina: ProSeRePEA Trial
Brief Title: Treatment of BPH With CO2 Serenoa +PEA as Monotherapy or in Combination With Tamsulosin: ProSeRePEA Trial
Acronym: ProSeRePEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Michele Billia, Medical doctor, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ProSeRePEA trial, v.01
Record Dates: First submitted 2022-04-08; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Benign Prostatic Hyperplasia; Urinary Obstruction; Lower Urinary Tract Symptoms
Keywords: BPH; benign prostatic hypertrophy
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The statistical analysis is blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ARM 1: PEAPROSTIL 600 mg + Tamsulosin 0.4 mg (Active Comparator): PEAPROSTIL 600 is a food supplement based on Palmitoylethanolamide and Serenoa Repens, respectively for each sachet there are 600 mg of PEA and 320 mg of Serenoa oil. The net content of a sachet is 2.45 g and can be orodispersible without the need for the use of water. The drug does not contain gluten or lactose.
  • Tamsulosin 0.4 mg is a drug belonging to the category of alpha-blocker drugs used as first choice drugs (according to European Urology association guidelines) for the treatment of LUTS/BPH. The recommended dose is 0.4 mg per day (1 administration), to be taken preferably at the same time during the day, indifferently with or without meals.
  Interventions: Drug: PEAPROSTIL 600 + Tamsulosin 0.4 mg
- ARM 2: PEAPROSTIL 600 mg (Active Comparator): PEAPROSTIL 600 is a food supplement based on Palmitoylethanolamide and Serenoa Repens, respectively for each sachet there are 600 mg of PEA and 320 mg of Serenoa oil. The net content of a sachet is 2.45 g and can be orodispersible without the need for the use of water. The drug does not contain gluten or lactose.
  Interventions: Drug: PEAPROSTIL 600 mg
- ARM 3: Tamsulosin 0.4 mg (Active Comparator): Tamsulosin 0.4 mg is a drug belonging to the category of alpha-blocker drugs used as first choice drugs (according to European Urology association guidelines) for the treatment of benign prostatic hyperplasia. The recommended dose is 0.4 mg per day (1 administration), to be taken preferably at the same time during the day, indifferently with or without meals.
  Interventions: Drug: Tamsulosin 0.4 mg

INTERVENTIONS:
Drug: PEAPROSTIL 600 + Tamsulosin 0.4 mg — PEAPROSTIL 600 mg one sachet oral daily+ Tamsulosin 0.4 mg one tablet oral daily
  Other Names: PEAPROSTIL, Omnic
  Arms: ARM 1: PEAPROSTIL 600 mg + Tamsulosin 0.4 mg
Drug: Tamsulosin 0.4 mg — Tamsulosin 0.4 mg one tablet oral daily
  Other Names: Omnic
  Arms: ARM 3: Tamsulosin 0.4 mg
Drug: PEAPROSTIL 600 mg — PEAPROSTIL 600 mg one sachet oral daily
  Other Names: PeaProstil
  Arms: ARM 2: PEAPROSTIL 600 mg

SUMMARY:
The objective of this study is to evaluate the efficacy of the supplement PEAPROSTIL 600 (FARMITALIA®) composed of Serenoa Repens combined with PEA in single or combined therapy with alpha-blocker in the reduction of voiding symptoms in benign prostatic hyperplasia (BPH) patients at low risk of progression to obstructing conditioning that need for surgical therapy. Any adverse events, intolerance, allergic reactions, complications related to the products used will be recorded throughout the study period.

DETAILED DESCRIPTION:
Study design

Single-center 3-arm randomized prospective clinical trial.

* Arm 1: PEAPROSTIL 600 + Tamsulosin 0.4 mg
* Arm 2: PEAPROSTIL 600
* Arm 3: Tamsulosin 0.4 mg

At the time of study enrollment, each patient will be randomized into one of the 3 arms described. Randomisation will take place with a 1: 1: 1 scheme.

All the variables will be collected by a medical co-investigator of Prof. Alessandro Volpe's team during the follow-up visits at pre-established intervals of 1, 3, 6 and 12 months (respectively T1, T2, T3 and T4) and will be reported in the special data collection folder (CRF).

At 1 month (T1) 3 months (T2), 6 months (T3) and 12 months (T4):

Personal data: identification number and initials of the patient's name and surname, date of birth, telephone number and e-mail address History: International Prostate Symptoms Score questionnaire, Short Form Health Survey-36 questionnaires Physical examination: abdominal, urological including rectal examination Uroflowmetry: analysis of the morphology of the flow curve, Qmax, volume of urine emptied, post-voiding residue).

250 patients will be recruited. The sample analysis was performed by the Department of Medical, Surgical and Advanced Technologies "Ingrassia" of the University of Catania for a study power of 90% and an Alpha error of 0.05 (statistical significance). In particular, the design involves a 3-arm randomization process 1: 1: 1. Expecting a difference of at least 2 points in the International Prostate Symptoms Score questionnaire and Qmax and a standard deviation of 4. It is necessary to enroll 250 patients to obtain a statistic of 90% at a significance level of 0.05. The statistical analysis of the data collected during the study, according to an intention-to-treat procedure, will be performed using statistical software including IBM SPSS statistics version 23.0. A descriptive analysis of the patients included in the three arms will be performed using the appropriate frequency measurements and central tendency and dispersion indices. Considering a pair of the three arms at a time (1 vs. 2; 1 vs. 3; 2 vs. 3), the qualitative variables will be compared using the chi-squared test; quantitative variables will be compared by Student's t-test. The significance level will be set at p <0.05. For the variables that will be significant in the univariate analysis, multivariate analyzes will be carried out using appropriate regression models.

ELIGIBILITY:
Inclusion Criteria:

* male with age> 40 years
* baseline International Prostate Symptoms Score between 8 and 14
* prostate volume ≤ 60 cc assessed by transrectal ultrasound (TRUS)
* maximum flow (Qmax at uroflowmetry) ≤ 15 ml / sec
* post voiding residue on extemporaneous ultrasound ≤ 120 ml
* Signature of informed consent for participation in the study
* ability to understand the conditions of the study and to participate in the study throughout its duration.

Exclusion Criteria:

* urinary incontinence
* overactive bladder
* neurological bladder
* malignancies in progress and which have undergone treatment in the previous 6 months
* local or systemic infections (urinary tract infection, osteomyelitis, sepsis, etc.)
* kidney failure
* macrohematuria
* bladder stones

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment of combination therapy group vs tamsulosin group in International Prostate Symptoms Score questionnaire | 1 year
  comparing patients receiving tamsulosin + peaprostil combination therapy (Arm 1) versus patients receiving tamsulosin monotherapy (Arm 3) in terms of International Prostate Symptoms Score (scale 0-35) at 1,3,6 and 12 months.
  (0 point no symptoms, 35 points many symptoms)
Efficacy of treatment of combination therapy group vs tamsulosin group in Quality of Life questionnaire | 1 year
  comparing patients receiving tamsulosin + peaprostil combination therapy (Arm 1) versus patients receiving tamsulosin monotherapy (Arm 3) in terms of Quality of life (0-6 points) at 1,3,6 and 12 months (0 point good quality of life, 6 points bad quality of life)

SECONDARY OUTCOMES:
Efficacy of treatment in combination therapy group vs tamsulosin group in evaluation of Short Form Health Survey-36 questionnaires | 1 year
  comparing patients receiving tamsulosin + peaprostil combination therapy (Arm 1) versus patients receiving tamsulosin monotherapy (Arm 3) in terms of Short Form Health Survey-36 (36 questions) at 1,3,6 and 12 months
Efficacy of treatment in combination therapy group vs tamsulosin group in evaluation of uroflowmetry with maximum urinary flow (ml/s) | 1 year
  comparing patients receiving tamsulosin + peaprostil combination therapy (Arm 1) versus patients receiving tamsulosin monotherapy (Arm 3) in terms of maximum urinary flow (ml/s) at 1,3,6 and 12 months
Efficacy of treatment in combination therapy group vs tamsulosin group in evaluation of post voided volume (ml) | 1 year
  comparing patients receiving tamsulosin + peaprostil combination therapy (Arm 1) versus patients receiving tamsulosin monotherapy (Arm 3) in terms of post voided volume (ml) at 1,3,6 and 12 months
Efficacy of treatment in combination therapy group vs tamsulosin group in evaluation of prostate volume (gr) | 1 year
  comparing patients receiving tamsulosin + peaprostil combination therapy (Arm 1) versus patients receiving tamsulosin monotherapy (Arm 3) in terms of prostate volume (gr) at 6 and 12 months
Efficacy of treatment in combination therapy group vs peaprostil group and peaprostil group vs tamsulosin group in terms of International Prostate Symptoms Score | 1 year
  comparing patients receiving combination therapy group (Arm1) vs peaprostil group (Arm2) and peaprostil group (Arm2) vs tamsulosin alone (Arm 3) in terms of International Prostate Symptoms Score (scale 0-35) at 1,3,6 and 12 months.
  (0 point no symptoms, 35 points many symptoms)
Efficacy of treatment in combination therapy group vs peaprostil group and peaprostil group vs tamsulosin group in terms of Quality of life | 1 year
  comparing patients receiving combination therapy group (Arm1) vs peaprostil group (Arm2) and peaprostil group (Arm2) vs tamsulosin alone (Arm 3) in terms of Quality of life (QoL) (0-6 points) at 1,3,6 and 12 months (0 point good quality of life, 6 points bad quality of life)
Efficacy of treatment in combination therapy group vs peaprostil group and peaprostil group vs tamsulosin group in terms of Short Form Health Survey-36 questionnaires | 1 year
  comparing patients receiving combination therapy group (Arm1) vs peaprostil group (Arm2) and peaprostil group (Arm2) vs tamsulosin alone (Arm 3) in terms of Short Form Health Survey-36 (36 questions) at 1,3,6 and 12 months
Efficacy of treatment in combination therapy group vs peaprostil group and peaprostil group vs tamsulosin group in terms of uroflowmetry with maximum urinary flow (ml/s) | 1 year
  comparing patients receiving combination therapy group (Arm1) vs peaprostil group (Arm2) and peaprostil group (Arm2) vs tamsulosin alone (Arm 3) in terms of maximum urinary flow (ml/s) at 1,3,6 and 12 months
Efficacy of treatment in combination therapy group vs peaprostil group and peaprostil group vs tamsulosin group in terms of post voided volume (ml) | 1 year
  comparing patients receiving combination therapy group (Arm1) vs peaprostil group (Arm2) and peaprostil group (Arm2) vs tamsulosin alone (Arm 3) in terms of post voided volume (ml) at 1,3,6 and 12 months
Efficacy of treatment in combination therapy group vs peaprostil group and peaprostil group vs tamsulosin group in terms of prostate volume (gr) | 1 year
  comparing patients receiving combination therapy group (Arm1) vs peaprostil group (Arm2) and peaprostil group (Arm2) vs tamsulosin alone (Arm 3) in terms of prostate volume (gr) at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michele Billia, MD, Principal Investigator — SCDU Urologia
Locations (1):
- Michele Billia, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT06181175/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT06181175/ICF_001.pdf